CLINICAL TRIAL: NCT05037188
Title: A Randomized, Double-blind, Placebo-controlled, Adaptive, Seamless Phase I / II Clinical Study of the Safety and Immunogenicity of a Recombinant Viral Vector AAV5-RBD-S Vaccine for the Prevention of Coronavirus Infection (COVID-19)
Brief Title: Clinical Study of the Safety and Immunogenicity of a Recombinant Viral Vector AAV5 (Adeno-Associated Virus Type 5 )-RBD (Receptor Binding Domain)-S Vaccine for the Prevention of Coronavirus Infection (COVID-19)
Acronym: COVER
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: BCD-250-1
Record Dates: First submitted 2021-09-07; First posted 2021-09-08 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection; COVID-19
Keywords: COVID-19 Vaccine; COVID-19 Virus Disease; COVID-19 Virus Infection; SARS-CoV-2 Infection
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Stage 1. Subjects without history of COVID-19 infection will be randomized in two treatment groups to receive different doses of BCD-250. After the last subject completes the 28 days of the main study period the safety and immunogenicity analysis will be performed. Based on these results the optimal BCD-250 dose will be selected by the Sponsor considering the Independent Data Monitoring Committee recommendations.
  Stage 2. Subjects without history of COVID-19 infection (Cohort 1) and with history of COVID-19 infection (Cohort 2) will be randomized to receive either selected dose of BCD-250 or placebo.
Who Masked: Participant, Investigator
Masking Description: Stage 1 will be open label. The participants will receive the assigned dose of BCD-250 according to the allocation.
  Stage 2 will be double blind, placebo-controlled. Investigators and subjects will be unaware of the assigned treatment (BCD-250 or placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- COVID-19 vaccine candidate (BCD-250) low dose (Experimental): The participants will receive the low dose of BCD-250
  Interventions: Biological: Low dose BCD-250 injection
- COVID-19 vaccine candidate (BCD-250) high dose (Experimental): The participants will receive the high dose of BCD-250
  Interventions: Biological: High dose BCD-250 injection
- Cohort 1/COVID-19 vaccine candidate (BCD-250) (Experimental): The participants will receive the selected dose of BCD-250
  Interventions: Biological: Low dose or high dose BCD-250 injection
- Cohort 1/Placebo (Placebo Comparator): The participants will receive placebo
  Interventions: Other: Placebo injection
- Cohort 2/COVID-19 vaccine candidate (BCD-250) (Experimental): The participants will receive the selected dose of BCD-250
  Interventions: Biological: Low dose or high dose BCD-250 injection
- Cohort 2/Placebo (Placebo Comparator): The participants will receive placebo
  Interventions: Other: Placebo injection

INTERVENTIONS:
Biological: Low dose BCD-250 injection — A recombinant viral vector AAV5-RBD-S vaccine
  Arms: COVID-19 vaccine candidate (BCD-250) low dose
Biological: High dose BCD-250 injection — A recombinant viral vector AAV5-RBD-S vaccine
  Arms: COVID-19 vaccine candidate (BCD-250) high dose
Biological: Low dose or high dose BCD-250 injection — A recombinant viral vector AAV5-RBD-S vaccine
  Arms: Cohort 1/COVID-19 vaccine candidate (BCD-250); Cohort 2/COVID-19 vaccine candidate (BCD-250)
Other: Placebo injection — Placebo injection
  Arms: Cohort 1/Placebo; Cohort 2/Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, adaptive, seamless phase I / II clinical study of the safety and immunogenicity of a recombinant viral vector AAV5-RBD-S vaccine for the prevention of coronavirus infection (COVID-19)

DETAILED DESCRIPTION:
The study will be carried out in 2 stages. Stage 1 aims to assess the safety and immunogenicity of different doses of BCD-250 in subjects without a history of COVID-19 infection to choose the optimal dose for further investigation.

Stage 2 aims to assess the immunogenicity and safety of the chosen on stage 1 optimal BCD-250 dose compared to placebo in subjects with and without the history of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Ability to comply with the study procedures based on the Investigator's assessment
* Males and females aged 18-60 years, inclusive, at the date of consent.
* Negative pregnancy test (for females of childbearing potential)
* Patients of childbearing potential and their partners with preserved reproductive function must agree to use reliable contraceptive methods starting from the time of informed consent for 3 months after Visit 1. This requirement does not apply to patients and their partners who underwent surgical sterilization. Reliable contraceptive methods include one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives.
* Cohort 1 only. Negative test for SARS-CoV-2 IgM and IgG at screening
* Cohort 2 only. Negative test for SARS-CoV-2 IgM at screening
* Cohort 2 only. Confirmed by SARS-CoV-2 RNA test, history of COVID-19 with documented recovery at least 4 month prior consent date.

Exclusion Criteria:

* Positive / uncertain test for SARS-CoV-2 RNA at screening
* Cohort 1 only. Documented history of COVID-19.
* Changes on chest X-ray suggestive for pneumonia or other lung diseases at screening, excluding clinically non-significant changes in subjects with COVID-19 history on investigator's opinion.
* Prior administration of SARS-CoV-2 or other coronavirus vaccine or planning of receiving SARS-CoV-2 or other coronavirus vaccine during the study participation.
* Known contact with SARS-CoV-2 infected person or person with known contact with SARS-CoV-2 infected person, within 14 days prior to consent date.
* Any acute infectious or non-infectious disease, including convalescence period, less than 4 weeks since clinical recovery
* Positive HIV, HBV, HCV or Syphilis tests
* History of splenectomy
* History of severe allergic reactions
* History of allergic or postvaccinal reactions (anaphylactic shock, fever of 40°C or more, fainting, non-febrile convulsions etc.) after vaccine administration
* Suspicious hypersensitivity or history of hypersensitivity to any component of investigational product
* Participation in other clinical studies within 90 days prior to consent date, excluding screen failures or discontinued prior to the first investigational product administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG titer from baseline | Day 56 after the study drug administration
  Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG titer (binding and neutralizing) from baseline on Day 56

SECONDARY OUTCOMES:
Percentage of subjects with acute immediate hypersensitivity reactions | 30 minutes after the study drug administration
  Percentage of subjects with acute immediate hypersensitivity reactions developed within 30 minutes after study drug administration.
Percentage of subjects with solicited local adverse reactions | 7 days after the study drug administration
  Percentage of subjects with local post-vaccination reactions developed within 7 days after study drug administration.
Percentage of subjects with grade ≥3 solicited local adverse reactions | 7 days after the study drug administration
  Percentage of subjects with grade ≥3 local post-vaccination reactions developed within 7 days after study drug administration.
Percentage of subjects with solicited systemic adverse reactions | 7 days after the study drug administration
  Percentage of subjects with systemic post-vaccination reactions developed within 7 days of study drug administration.
Percentage of subjects with grade ≥3 solicited systemic adverse reactions | 7 days after the study drug administration
  Percentage of subjects with grade ≥3 systemic post-vaccination reactions developed within 7 days of study drug administration.
Percentage of subjects with any adverse reactions | 56 days after the study drug administration
  Percentage of subjects with any adverse reactions developed within 56 days of study drug administration.
Percentage of subjects with any grade ≥3 adverse reactions | 56 days after the study drug administration
  Percentage of subjects with any grade ≥3 adverse reactions developed within 56 days of study drug administration.
The proportion of subjects with clinical and laboratory abnormalities | 56 days after the study drug administration
  The proportion of subjects with clinical and laboratory abnormalities developed within 56 days after administration of the study drug
Percentage of subjects with adverse events of special interest | up to Day 365
  Adverse events of special interest include the following adverse events: 1) AEs demanding the medical care, 2) Newly developed chronic diseases, 3) serious adverse reactions 4) Laboratory confirmed COVID-19 cases
Percentage of subjects with SARS-CoV-2-specific IgG antibodies | Days 7, 14, 21, 28, 56 after the study drug administration.
  Percentage of subjects with SARS-CoV-2-specific IgG (binding and neutralizing) antibodies within the main period of the study
Geometric mean titer of SARS-CoV-2-specific IgG antibodies | Days 7, 14, 21, 28, 56 after the study drug administration
  Geometric mean titer of SARS-CoV-2-specific IgG (binding and neutralizing) antibodies within the main period of the study
Change of the SARS-CoV-2-specific IgG antibodies titer from baseline | Days 7, 14, 21, 28, 56 after the study drug administration
  Change of the SARS-CoV-2-specific IgG (binding and neutralizing) antibodies titer from baseline within the main period of the study
Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG antibodies titer from baseline | Days 7, 14, 21, 28 after the study drug administration
  Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG (binding and neutralizing) antibodies titer from baseline within the main period of the study
Percentage of subjects with detected SARS-CoV-2-specific peripheral blood lymphocytes | Days 14, 28, 56 after the study drug administration.
  Percentage of subjects with detected SARS-CoV-2-specific peripheral blood lymphocytes within the main period of the study
Mean change in SARS-CoV-2-specific peripheral blood lymphocytes count | Days 14, 28, 56 after the study drug administration
  Mean change in SARS-CoV-2-specific peripheral blood lymphocytes count within the main period of the study
Percentage of subjects with SARS-CoV-2-specific IgG antibodies | Days 57- 365
  Percentage of subjects with SARS-CoV-2-specific IgG (binding and neutralizing) antibodies during the study
Geometric mean titer of SARS-CoV-2-specific IgG antibodies | Days 57- 365
  Geometric mean titer of SARS-CoV-2-specific IgG (binding and neutralizing) antibodies during the study
Change in the SARS-CoV-2-specific IgG titer from baseline | Days 57- 365
  Change in the SARS-CoV-2-specific IgG (binding and neutralizing) antibodies titer from baseline during the study
Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG (binding and neutralizing) titer from baseline | Days 57- 365
  Percentage of subjects with ≥ 4 fold rise of serum SARS-CoV-2-specific IgG titer from baseline during the study

OTHER OUTCOMES:
The proportion of subjects with identified AAV5 in biological fluids (blood, saliva and urine) | up to Day 365
  The proportion of subjects with identified AAV5 in biological fluids (blood, saliva and urine) during the study
Percentage of subjects with AAV5-specific IgG antibodies | up to Day 365
  Percentage of subjects with AAV5-specific IgG antibodies during the study

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - UNINOVA clinic, Saint Petersburg
  - X7 Clinical Research, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No